CLINICAL TRIAL: NCT06870279
Title: A Clinical Research Evaluating the Safety and Efficacy of CD70-targeted CAR-NKT Cells (CGC738) Therapy in Subjects With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: A Clinical Research of CD70-targeted CAR-NKT Cells (CGC738) Therapy in RCC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC738-IIT-02
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NKT Cells Lymphodepleting regimen (Experimental): CAR-NKT Cells treatment
  Interventions: Drug: CGC738

INTERVENTIONS:
Drug: CGC738 — CAR-NKT Cells treatment

SUMMARY:
This is a phase I, open-label, single-arm study conducted to evaluate the efficacy, safety and PK of CGC738 in the treatment of advanced clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
This is a single-arm, open-label study. This study will include two parts, dose escalation phase (3+3 design) followed by a dose expansion phase. All eligible participants will receive a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by CAR-T cell injection.

Additional patients will be enrolled in the dose expansion phase to further characterize the safety profile and evaluate the efficacy of anti-CD70 CAR-T cell injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 75 years.
* 2.ECOG 0-1 points.
* 3. The expected survival time is more than 3 months.
* 4. Patients with advanced ccRCC confirmed by histology or cytology to be recurrent or metastatic after at least first-line treatment.
* 5. IHC: CD70 positive.
* 6. At least one measurable lesion at baseline per RECIST version 1.1.
* 7. The functions of important organs are basically normal:
* 8. Pregnancy tests for women of childbearing age shall be negative, both men and women agreed to use effective contraception.

Exclusion Criteria:

* 1. Use of cell therapy within the previous one month.
* 2. Subjects with other malignant tumors within the past 2 years, except basal or squamous skin cancer, superficial bladder cancer, and breast cancer in situ, have been completely cured and do not need follow-up treatment.
* 3. Patients with leptomeningeal metastasis or central nervous system metastasis, and definite central nervous system underlying diseases with significant symptoms.
* 4. Immunotherapy, targeted drug therapy or chemotherapy within 5 drug half-lives within 2 weeks before cell infusion.
* 5. Active hepatitis B, HIV positive and HCV positive.
* 6. Active infection or uncontrollable infection.
* 7. Uncontrollable or significant heart disease.
* 8. Unstable respiratory diseases, including interstitial pneumonia.
* 9. Uncontrolled ascites and pleural effusion.
* 10.Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, etc.
* 11.Subjects who are using systemic steroids or steroid inhalers for treatment.
* 12.Pregnant or lactating female subjects.
* 13.Other investigators deem it unsuitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) | Day 28 after CGC738 infusion
  Dose limiting toxicity (DLT) is an AE that meets the following criteria and occurs within 28 days of CGC738 infusion.AE is graded according to CTCAE version 5.0.

SECONDARY OUTCOMES:
ORR | Day 1 through week 56
  Assess Objective response rate
DCR | Day 1 through week 56
  Assess Disease control rate
AEs | Day 1 through week 56
  Incidence of adverse events